CLINICAL TRIAL: NCT07192549
Title: Perioperative GDNF as a Predictive Factor for Postoperative Delirium and Adverse Neurological Outcomes in Pediatric Surgery:a Single-center, Prospective, Randomized Controlled Study
Brief Title: Perioperative GDNF as a Predictive Factor for Postoperative Delirium and Adverse Neurological Outcomes in Pediatric Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hui Wang-2025.9
Record Dates: First submitted 2025-09-10; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Delirium
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane Group (Experimental): Anesthesia was maintained with sevoflurane (Inhalation Sevoflurane, Brand: Kaiteli, Specification: 120 mL, Approval Number: National Drug Approval H20070172, Manufacturer: Shanghai Hengrui Pharmaceutical) combined with continuous intravenous infusion of remifentanil.
  Interventions: Drug: Sevoflurane group
- Propofol Group (Active Comparator): Anesthesia was maintained with remifentanil combined with continuous intravenous infusion of propofol at a maintenance dose of 0.5 mg/(kg·h).
  Interventions: Drug: Propofol group

INTERVENTIONS:
Drug: Sevoflurane group — Patients fasted for 6 hours and abstained from clear fluids for 3 hours preoperatively. Upon entering the operating room, oxygen was administered via an appropriately sized face mask at a flow rate of 6-8 L/min. Anesthesia was induced by sequential intravenous injection of remimazolam, sufentanil, and rocuronium. A laryngeal mask was inserted after the disappearance of the eyelash reflex. Anesthesia was maintained with sevoflurane (Inhalation Sevoflurane, Brand: Kaiteli, Specification: 120 mL, Approval Number: National Drug Approval H20070172, Manufacturer: Shanghai Hengrui Pharmaceutical) combined with continuous intravenous infusion of remifentanil. During surgery, vital signs and body movement responses were closely monitored, and the inhaled concentration of sevoflurane was adjusted as needed (maintained at 1%-3%). Administration of anesthetics was discontinued 5 minutes before the end of surgery.
  Arms: Sevoflurane Group
Drug: Propofol group — Preoperative preparation was identical to that of the Sevoflurane Group. Anesthesia induction was performed using the same sequence of intravenous injections of remimazolam, sufentanil, and rocuronium, followed by laryngeal mask insertion after the disappearance of the eyelash reflex. Anesthesia was maintained with remifentanil combined with continuous intravenous infusion of propofol at a maintenance dose of 0.5 mg/(kg·h). The infusion rate was dynamically adjusted based on intraoperative vital signs. Administration of anesthetics was stopped 5 minutes before the end of surgery.
  Arms: Propofol Group

SUMMARY:
To observe the dynamic changes in serum levels of inflammatory cytokines (e.g., IL-6, TNF-α), Brain-Derived Neurotrophic Factor (BDNF), and Glial Cell Line-Derived Neurotrophic Factor (GDNF) during the perioperative period in pediatric patients undergoing Scheduled Laparoscopic Hernia Repair surgery, and to investigate their relationship with the occurrence of postoperative delirium (POD) and postoperative cognitive dysfunction (POCD),and to compare the different influence between propofol and sevoflurane . The aim is to provide insights into the neurobiological mechanisms underlying these complications and to identify potential biomarkers for risk stratification.

DETAILED DESCRIPTION:
Clarify the Correlation Between Perioperative Changes in Inflammatory Factors, BDNF, and GDNF Levels and Postoperative delirium (POD) Blood and urine samples were collected from pediatric patients at three time points: 5 minutes before anesthesia induction (T0), 1 hour after surgery began (T1), and on the first postoperative day (T2). Serum levels of inflammatory factors (such as IL-6 and TNF-α) as well as brain-derived neurotrophic factor (BDNF) and glial cell line-derived neurotrophic factor (GDNF) were measured. The Richmond Agitation-Sedation Scale (RASS) was used to assess the children within 5-10 minutes after awakening from anesthesia. The RASS score ranges from +4 (combative agitation) to -5 (coma), comprising 10 levels, with higher scores indicating more agitated states and lower scores indicating deeper sedation. A score ≥+1 was defined as agitation. By comparing changes in inflammatory factors and neurotrophic factor levels across different time points, the association with the occurrence of postoperative agitation was analyzed.

Clarify the Correlation Between Perioperative Changes in Inflammatory Factors, BDNF, and GDNF Levels and Learning and Memory Abilities at Age 5 For the same cohort of children, based on blood and urine samples collected at the aforementioned time points (T0, T1, T2), concentrations of inflammatory factors (such as IL-6 and TNF-α), BDNF, and GDNF were measured. When the children reached 5 years of age, standardized neurocognitive assessment tools (such as the Wechsler Preschool and Primary Scale of Intelligence-IV [WPPSI-IV] or age-appropriate memory and learning function tests) were used to evaluate their learning and memory abilities. Statistical analysis was performed to explore the potential correlation between the dynamic changes in the aforementioned biomarkers during the perioperative period and cognitive function scores at age 5.

ELIGIBILITY:
Inclusion Criteria:

* (1) Aged 1-3 years; (2) American Society of Anesthesiologists (ASA) Physical Status Classification I-II; (3) Body Mass Index (BMI) 18-35 kg/m²; (4) Agreement to participate in the study and signed informed consent form.

Exclusion Criteria:

* (1) Surgical duration exceeding 4 hours; (2) Patients with language or hearing impairments hindering effective communication; (3) Patients with postoperative infections or perioperative cardiopulmonary complications; (4) Patients with preoperative psychiatric disorders.

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between Perioperative Inflammatory Factors and Neurotrophic Factor Levels with Postoperative Delirium | Preoperative to postoperative day 1
  The levels of inflammatory factors IL-1β, IL-6, and TNF-α in pediatric patients will be measured using ELISA before surgery, 30 minutes during surgery, and one day after surgery. Simultaneously, the levels of neurotrophic factors BDNF and GDNF will be detected using ELISA. The RASS scale was employed to assess the level of emergence agitation in the children. A t-test will be used to compare whether the inflammatory factor levels between the two groups were correlated with the occurrence of emergence agitation, to determine whether the pre- and postoperative changes in neurotrophic factors are statistically significant, and to evaluate whether these changes is correlated with the incidence of emergence agitation.
Correlation between Perioperative Inflammatory Factors and Neurotrophic Factor Levels with Neurodevelopmental Outcomes at 5 Years of Age | Preoperative until the child reaches 5 years of age
  The levels of inflammatory factors IL-1β, IL-6, and TNF-α in pediatric patients will be measured using ELISA before surgery, 30 minutes during surgery, and one day after surgery. Simultaneously, the levels of neurotrophic factors BDNF and GDNF will be detected using ELISA. The Wechsler Scale II will be employed to assess the learning and memory abilities of the children at five years of age. A t-test was used to compare whether the inflammatory factor levels between the two groups will be correlated with the development of long-term learning and memory function, and to evaluate whether changes in these levels were associated with the occurrence of long-term learning and memory function.

SECONDARY OUTCOMES:
Correlation between Surgical Type on the Expression of Inflammatory Factors with Neurotrophic Factors | Intraoperative to postoperative day 1
  We will categorize the surgeries into upper abdominal, lower abdominal, and limb procedures based on human anatomical structure. Correlation analysis will performe between these surgical categories and the levels of inflammatory factors and neurotrophic factors measured by ELISA. This analysis aim to evaluate whether the type of surgery will correlate with changes in inflammatory factor levels, as well as to examine the association between surgical categories and the occurrence of postoperative delirium.
Correlation between Surgical Duration on the Expression of Inflammatory Factors with Neurotrophic Factors | Intraoperative to postoperative day 1
  We will classify the surgeries into two categories based on a 2-hour duration threshold and performed correlation analysis with the levels of inflammatory factors and neurotrophic factors measured by ELISA. This analysis aimed to evaluate whether the duration of surgery was correlated with changes in inflammatory factor levels, as well as to examine the association between surgical duration and the occurrence of emergence delirium and long-term neurological function.
Collection between Anesthetic Drugs on the Expression of Inflammatory Factors with Neurotrophic Factors | Intraoperative to postoperative day 1
  We will categorize the surgeries into propofol-based maintenance group and sevoflurane-based maintenance group. Correlation analysis will be performed between these two anesthetic approaches and the levels of inflammatory factors and neurotrophic factors measured by ELISA. This analysis aim to evaluate whether the choice of anesthetic agent was correlated with alterations in inflammatory factor levels.